CLINICAL TRIAL: NCT06195488
Title: Preoperative Evaluation of Gastric Contents in Diabetic Patients With Gastric Ultrasound
Brief Title: Gastric Ultrasound in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bengü Gülhan Köksal, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2022/17-1
Record Dates: First submitted 2023-11-24; First posted 2024-01-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gastric Emptying; Diabetes; Ultrasound
Keywords: fasting; gastric ultrasound; preoperative fasting; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group D: Group Diabetic
  Interventions: Procedure: Gastric ultrasound
- Group Control: Non-diabetic patients
  Interventions: Procedure: Gastric ultrasound

INTERVENTIONS:
Procedure: Gastric ultrasound — performing gastric ultrasound to determine gastric contents

SUMMARY:
The American Society of Anesthesiologists (ASA) does not specify a fasting period for patients with certain comorbidities, such as diabetes, for elective surgery, and does not make a separate recommendation for surgery.

The European Society of Anesthesiology (ESA) guidelines do not differentiate between diabetic patients and normal patients. Aspiration of gastric contents is a common cause of perioperative morbidity and mortality.

Aspiration can cause hypoxia, bronchospasm, pneumonia, acute respiratory distress syndrome and death.

The presence of food or fluid in the stomach before induction of anesthesia is one of the greatest risk factors for perioperative pulmonary aspiration. Sedation and general anesthesia suppress or inhibit physiologic mechanisms (tone of the lower esophageal sphincter and upper airway reflexes) that protect against aspiration.

Because restriction of fluid and food intake before general anesthesia is vital for patient safety, Anesthesiology societies have developed guidelines for preoperative fasting.

Current ASA guidelines recommend at least 2 hours fasting for clear liquids, 6 hours fasting after a light meal (toast and clear liquids) and 8 hours fasting after a high calorie or fat meal. The information obtained from gastric ultrasound allows anesthesiologists to determine the optimal timing of procedures, type of anesthesia and airway management technique.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained 40-65 BMI<40 ASA I-III Fasting for at least 8 hours Elective surgery

Exclusion Criteria:

* Pregnancy Upper gastrointestinal malignancy Large Hiatal Hernia Kidney failure Liver failure Opioid use Use of drugs affecting motility Previous upper abdominal surgery BMI ≥40 kg/m2 Emergency surgery Diabetic ketoacidosis Sepsis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic and non-diabetic patients aged 40-65 years undergoing ASA I-III elective surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
determine stomach fullness | baseline (before intubation)
  To evaluate residual gastric volume in diabetic patients fasting for elective surgery

SECONDARY OUTCOMES:
Incidence of risk factors | during surgery
  Investigating risk factors for a full stomach in diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No